CLINICAL TRIAL: NCT00972881
Title: EXCITE: Erbitux, Xeloda, Campto, Irradiation Then Excision for Locally Advanced Rectal Cancer (North West Clinical Oncology Group-04 on Behalf of the NCRI Rectal Cancer Subgroup)
Brief Title: Capecitabine, Irinotecan Hydrochloride, Cetuximab, and Radiation Therapy in Treating Patients Undergoing Surgery for Locally Advanced Rectal Cancer
Acronym: EXCITE
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University College, London (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000648171; CRUK-UCL-EXCITE; EUDRACT-2007-006701-25; EU-20964
Record Dates: First submitted 2009-09-05; First posted 2009-09-09 (Estimated); Last update posted 2017-10-25 (Actual); Status verified 2014-12

CONDITIONS: Rectal Cancer
Keywords: adenocarcinoma of the rectum; Locally advanced rectal cancer
MeSH Terms: conditions — Rectal Neoplasms | interventions — Cetuximab; Capecitabine; Irinotecan; Neoadjuvant Therapy; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Biological: cetuximab
Drug: capecitabine
Drug: irinotecan hydrochloride
Procedure: neoadjuvant therapy
Procedure: therapeutic conventional surgery
Radiation: radiation therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as capecitabine and irinotecan hydrochloride, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Monoclonal antibodies, such as cetuximab, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them. Radiation therapy uses high-energy x-rays to kill tumor cells. Giving combination chemotherapy, cetuximab, and radiation therapy before surgery may make the tumor smaller and reduce the amount of normal tissue that needs to be removed.

PURPOSE: This phase I/II trial is studying the side effects of giving capecitabine and irinotecan hydrochloride together with cetuximab and radiation therapy and to see how well it works in treating patients undergoing surgery for locally advanced rectal cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* To assess the downstaging effectiveness and tolerability of neoadjuvant chemoradiotherapy comprising capecitabine, irinotecan hydrochloride, cetuximab, and radiotherapy in patients with locally advanced rectal cancer.

OUTLINE: This is a multicenter study.

Patients receive cetuximab IV over 1-2 hours once weekly in weeks 1-6 and irinotecan hydrochloride IV over 1 hour once weekly in weeks 2-5. Patients also undergo pelvic radiotherapy once daily and receive oral capecitabine twice daily on days 1-5 in weeks 2-6.

Patients undergo surgery 8 weeks after completion of chemoradiotherapy.

After completion of study treatment, patients are followed up at 6, 12, 24, and 36 months.

Peer Reviewed and Funded or Endorsed by Cancer Research United Kindom (UK).

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed adenocarcinoma of the rectum
* MRI-defined locally advanced disease, as defined by 1 of the following:

  * Mesorectal fascia involvement
  * Mesorectal fascia threatened (tumor ≤ 1 mm from mesorectal fascia)
  * Any T3 tumor < 5 cm from anal verge
* No evidence of metastatic disease

PATIENT CHARACTERISTICS:

* ECOG or WHO performance status 0-1
* ANC ≥ 1.5 x 10^9/L
* Platelet count ≥ 100 x 10^9/L
* Serum bilirubin < 1.25 times upper limit of normal (ULN)
* Serum transaminase(s) < 3 times ULN
* Serum alkaline phosphatase < 5 times ULN
* Estimated glomerular filtration rate > 50 mL/min
* Not pregnant or nursing
* Fertile patients must use effective contraception
* Fit to receive all study treatments
* Able to comply with oral medication
* No comorbidity or coagulation problem that would deem the patient unsuitable for surgery
* No pre-existing condition that would preclude radiotherapy (e.g., fistulas, severe ulcerative colitis [particularly patients currently taking sulfasalazine], Crohn's disease, prior adhesions)
* No current or impending rectal obstruction (unless a defunctioning stoma is present) or metallic colonic rectal stent in situ
* No significant small bowel delineated within the radiotherapy fields
* No pelvic sepsis
* No gastrointestinal disorder that would interfere with oral therapy or oral bioavailability
* No uncontrolled cardiac, respiratory, or other disease that would preclude study therapy or informed consent
* No serious medical or psychiatric disorder that would preclude study therapy or informed consent
* No known dihydropyrimidine dehydrogenase deficiency

PRIOR CONCURRENT THERAPY:

* No prior chemotherapy
* No prior radiotherapy to the pelvis
* No concurrent participation in other studies, except genetic studies (e.g., NSCCG-National Study of Colorectal Cancer Genetics)
* No concurrent St. John wort
* No other concurrent cytotoxic treatment or radiotherapy

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2009-04; Primary Completion 2011-12 (Actual); Study Completion 2016-12-31 (Actual)

PRIMARY OUTCOMES:
Histologically confirmed R0 resection rate | Week 14 (6 weeks after treatment complete)

SECONDARY OUTCOMES:
Radiotherapy compliance | Weeks 2, 3, 4, 5 & 6
  Radiotherapy treatment and dosage is captured on weekly CRFs from week 2-6
Grade 3 or 4 toxicity as assessed by NCI CTCAE v3.0 | Baseline, week 1- 10, week 12 & 14 then at 6, 12, 24 & 36 months follow up
  Adverse events are recorded weekly on CRFs from week 1 of treatment until 4 weeks post treatment, then at 1 month post surgery and specified time points during long term follow up at 6, 12, 24 & 36 month intervals.
Pathological complete response | Week 14 (surgery conducted 6 weeks from end of treatment)
Post-operative morbidity | Week 14
Long-term morbidity | Week 14, then at 6, 12, 24 & 36 months follow up
Disease-free survival | Baseline, week 1- 10, week 12, 14 & then at 6, 12, 24 & 36 months follow up
Local failure-free survival | Baseline, weeks 1- 10, weeks 12 & 14 then at 6, 12, 24 & 36 months follow up

CONTACTS AND LOCATIONS:
Overall Officials: Simon Gollins, MD, Principal Investigator — Glan Clwyd Hospital
Locations (5):
- United Kingdom (5):
  - Yorkshire Regional Clinical Trials & Research Unit, Leeds, England
  - Christie Hospital, Manchester, England
  - Clatterbridge Centre for Oncology, Merseyside, England
  - Rosemere Cancer Centre at Royal Preston Hospital, Preston, England
  - Cancer Research UK and University College London Cancer Trials Centre, Rhyl, Denbighshire, Wales

REFERENCES:
- See also: Clinical trial summary from the Cancer Research UK website — http://www.cancerresearchuk.org/about-cancer/find-a-clinical-trial/a-trial-looking-at-cetuximab-capecitabine-and-irinotecan-with-radiotherapy-before-surgery-for-cancer-of-the-rectum